CLINICAL TRIAL: NCT07043491
Title: Comparison of Endoscopy and Esophagram for the Routine Evaluation of Anastomosis After McKeown Esophagectomy
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Professor, Sun Yat-sen University
Other Study IDs: B2024-656-01
Record Dates: First submitted 2025-06-02; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Cancer; Surgery-Complications
Keywords: Esophageal cancer; Endoscopy; Esophagram; McKeown esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopy group: The patients routinely underwent either endoscopy for the evaluation of anastomosis on postoperative day 7. The initiation of oral intake depended on the status of anastomosis according to the assessment result of endoscopy. The patients whose endoscopy revealed a good healing anastomosis were allowed to initiate oral intake. While the patients whose endoscopy revealed a poor healing anastomosis were monitored with a repeat endoscopy weekly and these patients were delayed for oral intake until the repeat endoscopy revealed a good healing anastomosis.
  Interventions: Diagnostic Test: Endoscopy
- Esophagram group: All patients routinely underwent esophagram for the evaluation of anastomosis on postoperative day 7. The initiation of oral intake depended on the status of anastomosis according to the assessment result of esophagram. The patients whose esophagram indicated an intact anastomosis were allowed to initiate oral intake.

INTERVENTIONS:
Diagnostic Test: Endoscopy — We first observed the residual esophagus to evaluate the mucosal color. We then reached the top of the anastomosis to obtain a full view of the anastomosis to exclude obvious leakage around that site. We next conducted a more detailed endoscopic examination at a close focal distance, circumferentially around the anastomosis. During this process, we utilized saline solution to meticulously remove white fibrin coverings and bloodstains to the greatest extent possible to ensure a thorough evaluation of anastomotic integrity. Finally, we inspected the staple line of the tubularized stomach to exclude gastric fistula and assessed the perfusion of the gastric graft. Endoscopic findings were assessed by an additional endoscopist and 3 esophageal surgeons during the examination, as well as by reviewing captured images or videos after endoscopy.
  Groups: Endoscopy group

SUMMARY:
This retrospective cohort study reviewed patients who underwent McKeown esophagectomy. All patients routinely underwent either endoscopy or esophagram for the evaluation of anastomosis on postoperative day 7. The initiation of oral intake depended on the status of anastomosis according to the assessment result of endoscopy or esophagram. All patients were followed up for six months after the assessment of anastomosis.

DETAILED DESCRIPTION:
This retrospective cohort study reviewed patients who underwent McKeown esophagectomy. All patients routinely underwent either endoscopy or esophagram for the evaluation of anastomosis on postoperative day 7. The initiation of oral intake depended on the status of anastomosis according to the assessment result of endoscopy or esophagram. The patients whose esophagram indicated an intact anastomosis or whose endoscopy revealed a good healing anastomosis were allowed to initiate oral intake. While the patients whose endoscopy revealed a poor healing anastomosis were monitored with a repeat endoscopy weekly and these patients were delayed for oral intake until the repeat endoscopy revealed a good healing anastomosis. All patients were followed up for six months after the assessment of anastomosis. The primary endpoints were the efficacy of the evaluation of anastomosis, which included the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) for AL, the accuracy of the evaluation of anastomosis, and the incidence of AL after oral intake. Cases of AL that were found after the previous assessment were regarded as missed diagnoses when the sensitivity was calculated. The secondary endpoints included the time from surgery to AL diagnosis, the time required for AL healing, and safety profile.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria required patients to have routinely undergone either endoscopy or an esophagram for the postoperative evaluation of anastomosis.

Exclusion Criteria:

We excluded the patient with histologically confirmed benign tumors of the esophagus or esophagogastric junction and the patient who had incomplete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study reviewed patients who underwent McKeown esophagectomy. All patients routinely underwent either endoscopy or esophagram for the evaluation of anastomosis on postoperative day 7.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-07-09 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The sensitivity for detecting AL | From January 1, 2022 to July 9, 2023
  The number of the patients who is true positive for AL/ The total number of AL
The specificity for detecting AL | From January 1, 2022 to July 9, 2023
  The number of the patients who is true negative for AL/ The total number of the patients who did not develop AL
Predictive positive value for AL | From January 1, 2022 to July 9, 2023
  The number of the patients who is true positive for AL/ The number of the patients who is evaluated as AL
Predictive negative value for AL | From January 1, 2022 to July 9, 2023
  The number of the patients who is true negative for AL/ The number of the patients who is determined to have an intact anastomosis
The incidence of AL after oral intake | From January 1, 2022 to July 9, 2023
  The number of the AL that occurs after oral intake/ The number of the patients who were determined to have an intact anastomosis

SECONDARY OUTCOMES:
The time from surgery to the diagnosis of AL | From January 1, 2022 to July 9, 2023
  The time from surgery to the diagnosis of AL
The time required for the healing of AL | From January 1, 2022 to July 9, 2023
  The degree of AL healing was determined on the basis of the evidence that no swallowed liquid flowed out of the anastomosis, accompanied by a repeat examination with a normal result and disappearance of clinical manifestations

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yang, PhD., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
It has not yet been determined